CLINICAL TRIAL: NCT03785379
Title: A Randomized Trial Evaluating the Effects of One-Year Caloric Restriction and 12-Week Exercise Training Intervention in Obese Adults With Type 2 Diabetes: Emphasis on Metabolic Control and Resting Metabolic Rate
Brief Title: A Trial Evaluating the Effects of a One-year Lifestyle Intervention in Obese Patients With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Padova (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2718P
Record Dates: First submitted 2018-10-26; First posted 2018-12-24 (Actual); Last update posted 2018-12-24 (Actual); Status verified 2018-12

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Obesity; Lifestyle intervention
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity | interventions — Caloric Restriction; Exercise

STUDY DESIGN:
Intervention Model Description: After the baseline assessment, patients will be randomly assigned either to: 1) 1-year caloric restriction with an immediate start of 12-week supervised structured exercise training (SSET) (Early-SSET intervention), followed by no exercise at health centers for 3 months; or: 2) 1-year caloric restriction with no exercise at health centers for 3 months and then a 12-week SSET from month 4 to month 6 (Late-SSET intervention). During the last 6 months participants' activity will be unrestricted.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Caloric restriction and early SSET (Active Comparator): Patients will participate to a short lifestyle intervention (LSI), consisting of four weekly group-led lessons lasting 60-90 minutes to educate them on specific dietary and physical activity recommendations for improving health and metabolic control. At the end of the 1-month LSI, participants will start a caloric restriction and early exercise training (SSET) during the first 12-week, followed by no exercise at health centers for 3 months. Between the 6- and the 12-month assessments, participants will continue caloric restriction and will be encouraged to freely exercise.
  Interventions: Behavioral: Caloric restriction; Behavioral: Exercise training
- Caloric restriction and late SSET (Active Comparator): Patients will participate to a short lifestyle intervention (LSI), consisting of four weekly group-led lessons lasting 60-90 minutes to educate them on specific dietary and physical activity recommendations for improving health and metabolic control. At the end of the 1-month LSI, participants will start a one-year caloric restriction with no exercise at health centers for 3 months, and then a 12-week exercise training (SSET). Between the 6- and the 12-month assessments, participants will continue caloric restriction and will be encouraged to freely exercise.
  Interventions: Behavioral: Caloric restriction; Behavioral: Exercise training

INTERVENTIONS:
Behavioral: Caloric restriction — A structured dietary training will be implemented to educate participants about recommended dietary habits.Patients will follow a caloric restriction (CR) diet, with an energy intake equal to the measured Resting Metabolic Rate (RMR) and with 45% carbohydrate, 20%protein, 35%fat, and 30 g/day fibers. At each follow-up, nutritionist will adjust CR to the latest measured RMR and assess the compliance to the diet.
  Other Names: One-year caloric restriction
Behavioral: Exercise training — Trainers will supervise participants during 12-weeks of structured exercise consisting of 150 min/week workouts, divided in three sessions of progressive mixed (aerobic and resistance) exercise. All aerobic exercise will be performed using treadmill and/or cycle ergo-meter.
  Other Names: 12-week structured supervised exercise training (SSET)

SUMMARY:
Diabetic patients with uncontrolled disease are often characterized by increased energy expenditure and could thus present a high resting metabolic rate (RMR). Lifestyle interventions aimed at improving glucose control in these patients may lead to reductions of futile pathways, resulting in lower rates of energy expenditure, and paradoxically to making it more difficult to lose weight. However, only few studies investigated how exercise could influence patients' RMR and results are still not unanimous. In this study, we aim to investigate the effects on metabolic health of a combined dietary intervention and 12-week exercise training in obese adults with type 2 diabetes.

DETAILED DESCRIPTION:
Although a number of exercise training interventions have been proposed to type 2 diabetes patients, the current clinical practice demonstrates that most patients are still sedentary and with excess body weight. A negative balance between energy intake and energy expenditure is crucial to reduce excess body weight. However, diabetic patients with uncontrolled disease are often characterized by increased energy expenditure and could thus present a high resting metabolic rate (RMR). Lifestyle interventions aimed at improving glucose control in these patients may lead to reductions of futile pathways, resulting in lower rates of energy expenditure, and paradoxically to making it more difficult to lose weight. However, no robust evidence has been collected on this issue, and the few studies that investigated how exercise could influence patients' RMR have not shown unanimous results, especially concerning combined dietary and physical activity interventions.

This open-label randomized trial in obese adults with type 2 diabetes aims to investigate the effects of a 1-year caloric restriction and 12-week exercise training intervention on metabolic health, RMR and VO2max.

In particular, eligible type 2 diabetes patients of our clinic will be invited to participate in a short lifestyle intervention (LSI). LSI will consist of four weekly group-led lessons lasting 60-90 minutes in which specialized professionals will educate patients on specific dietary and physical activity recommendations for improving health and metabolic control.

After this month, patients will be randomly assigned either to: 1) 1-year caloric restriction with an immediate start of 12-week supervised structured exercise training (SSET) (Early-SSET intervention), followed by no exercise at health centers for 3 months; or: 2) 1-year caloric restriction with no exercise at health centers for 3 months and then a 12-week SSET from month 4 to month 6 (Late-SSET intervention). During the last 6 months participants' activity will be unrestricted.

Type 2 diabetic and obese adult volunteers will be recruited and screened through medical history, physical examination and biochemical analyses.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* age 30 to 64 years
* less than 60 min aerobic exercise/week
* absence of acute diseases
* no current treatment with insulin or sulfonylureas

Exclusion Criteria:

* Body mass index (BMI)<28
* HbA1c<6%
* Recent acute diseases, severe infections, trauma or surgery
* Uncontrolled hypertension or hyperglycemia
* Evidence of advanced cardiovascular, renal or hepatic diseases
* Contraindication to exercise
* Body weight change of more than 3% within the last 6 months
* Medication changes within the last 3 months

Ages: 30 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline Glycated Hemoglobin (HbA1c) at 6 months | 6 months
  Venous blood samples will be collected at morning between 7-9 a.m. for the analysis of Glycated Hemoglobin, performed following standard quality-control procedures.

SECONDARY OUTCOMES:
Change from baseline Resting Metabolic Rate at 3 months | 3 months
  Resting Metabolic Rate will be measured using an open-circuit indirect calorimeter (Sensor Medics VO2max -229 Metabolic System, CA) under standardized procedures
Change from baseline Resting Metabolic Rate at 6 months | 6 months
  Resting Metabolic Rate will be measured using an open-circuit indirect calorimeter (Sensor Medics VO2max -229 Metabolic System, CA) under standardized procedures
Change from baseline Resting Metabolic Rate at 12 months | 12 months
  Resting Metabolic Rate will be measured using an open-circuit indirect calorimeter (Sensor Medics VO2max -229 Metabolic System, CA) under standardized procedures
Change from baseline Body mass index at 3 months | 3 months
  Body weight will be measured to the nearest 0.1 kg and height to the nearest 1 cm using a standard balance and stadiometer (Seca, Germany), with subjects wearing light clothing and no shoes. Body mass index will be computed from the ratio between weight (kg) and height (m) squared.
Change from baseline Body mass index at 6 months | 6 months
  Body weight will be measured to the nearest 0.1 kg and height to the nearest 1 cm using a standard balance and stadiometer (Seca, Germany), with subjects wearing light clothing and no shoes. Body mass index will be computed from the ratio between weight (kg) and height (m) squared.
Change from baseline Body mass index at 12 months | 12 months
  Body weight will be measured to the nearest 0.1 kg and height to the nearest 1 cm using a standard balance and stadiometer (Seca, Germany), with subjects wearing light clothing and no shoes. Body mass index will be computed from the ratio between weight (kg) and height (m) squared.
Change from baseline Fat-free mass at 3 months | 3 months
  Fat-free mass will be estimated by Dual Energy X-ray Absorptiometry, with fan-beam technology (Hologic QDR 4500 W, Inc.).
Change from baseline Fat-free mass at 6 months | 6 months
  Fat-free mass will be estimated by Dual Energy X-ray Absorptiometry, with fan-beam technology (Hologic QDR 4500 W, Inc.).
Change from baseline Fat-free mass at 12 months | 12 months
  Fat mass will be estimated by Dual Energy X-ray Absorptiometry, with fan-beam technology (Hologic QDR 4500 W, Inc.).
Change from baseline android to gynoid percent fat ratio at 3 months | 3 months
  Android to gynoid percent fat ratio will be estimated by Dual Energy X-ray Absorptiometry, with fan-beam technology (Hologic QDR 4500 W, Inc.).
Change from baseline android to gynoid percent fat ratio at 6 months | 6 months
  Android to gynoid percent fat ratio will be estimated by Dual Energy X-ray Absorptiometry, with fan-beam technology (Hologic QDR 4500 W, Inc.).
Change from baseline android to gynoid percent fat ratio at 12 months | 12 months
  Android to gynoid percent fat ratio will be estimated by Dual Energy X-ray Absorptiometry, with fan-beam technology (Hologic QDR 4500 W, Inc.).
Change from baseline fasting plasma glucose at 3 months | 3 months
  Venous blood samples will be collected in the morning between 7-9 a.m. after 12 hours of fasting and plasma glucose will be assessed following standard quality-control procedures.
Change from baseline fasting plasma glucose at 6 months | 6 months
  Venous blood samples will be collected in the morning between 7-9 a.m. after 12 hours of fasting and plasma glucose will be assessed following standard quality-control procedures.
Change from baseline fasting plasma glucose at 12 months | 12 months
  Venous blood samples will be collected in the morning between 7-9 a.m. after 12 hours of fasting and plasma glucose will be assessed following standard quality-control procedures.
Change from baseline HDL cholesterol at 3 months | 3 months
  Venous blood samples will be collected in the morning between 7-9 a.m. after 12 hours of fasting and HDL cholesterol will be assessed following standard quality-control procedures.
Change from baseline HDL cholesterol at 6 months | 6 months
  Venous blood samples will be collected in the morning between 7-9 a.m. after 12 hours of fasting and HDL cholesterol will be assessed following standard quality-control procedures.
Change from baseline HDL cholesterol at 12 months | 12 months
  Venous blood samples will be collected in the morning between 7-9 a.m. after 12 hours of fasting and HDL cholesterol will be assessed following standard quality-control procedures.
Change from baseline total cholesterol at 3 months | 3 months
  Venous blood samples will be collected in the morning between 7-9 a.m. after 12 hours of fasting and total cholesterol levels will be assessed following standard quality-control procedures.
Change from baseline total cholesterol at 6 months | 6 months
  Venous blood samples will be collected in the morning between 7-9 a.m. after 12 hours of fasting and total cholesterol levels will be assessed following standard quality-control procedures.
Change from baseline total cholesterol at 12 months | 12 months
  Venous blood samples will be collected in the morning between 7-9 a.m. after 12 hours of fasting and total cholesterol levels will be assessed following standard quality-control procedures.
Change from baseline triglycerides levels at 3 months | 3 months
  Venous blood samples will be collected in the morning between 7-9 a.m. after 12 hours of fasting and plasma triglycerides levels will be assessed following standard quality-control procedures.
Change from baseline triglycerides levels at 6 months | 6 months
  Venous blood samples will be collected in the morning between 7-9 a.m. after 12 hours of fasting and plasma triglycerides levels will be assessed following standard quality-control procedures.
Change from baseline triglycerides levels at 12 months | 12 months
  Venous blood samples will be collected in the morning between 7-9 a.m. after 12 hours of fasting and plasma triglycerides levels will be assessed following standard quality-control procedures.
Change from baseline serum creatinine at 3 months | 3 months
  Serum creatinine will be assessed from venous blood samples following standard quality-control procedures.
Change from baseline serum creatinine at 6 months | 6 months
  Serum creatinine will be assessed from venous blood samples following standard quality-control procedures.
Change from baseline serum creatinine at 12 months | 12 months
  Serum creatinine will be assessed from venous blood samples following standard quality-control procedures.
Change from baseline urinary albumin-to-creatinine ratio at 3 months | 3 months
  Urine samples will be collected for the assessment of urinary albumin-to-creatinine ratio (ACR) following standard quality-control procedures.
Change from baseline urinary albumin-to-creatinine ratio at 6 months | 6 months
  Urine samples will be collected for the assessment of urinary albumin-to-creatinine ratio (ACR) following standard quality-control procedures.
Change from baseline urinary albumin-to-creatinine ratio at 12 months | 12 months
  Urine samples will be collected for the assessment of urinary albumin-to-creatinine ratio (ACR) following standard quality-control procedures.
Change from baseline maximal aerobic power at 3 months | 3 months
  VO2max will be measured by the Sensor Medics VO2max -229 Metabolic System using a continuous incremental treadmill protocol (Runner MTC Climb, Italy) according to the modified Naughton protocol.
Change from baseline maximal aerobic power at 6 months | 6 months
  VO2max will be measured by the Sensor Medics VO2max -229 Metabolic System using a continuous incremental treadmill protocol (Runner MTC Climb, Italy) according to the modified Naughton protocol.
Change from baseline maximal aerobic power at 12 months | 12 months
  VO2max will be measured by the Sensor Medics VO2max -229 Metabolic System using a continuous incremental treadmill protocol (Runner MTC Climb, Italy) according to the modified Naughton protocol.
Change from baseline Glycated Hemoglobin (HbA1c) at 3 months | 3 months
  Venous blood samples will be collected at morning between 7-9 a.m. for the analysis of Glycated Hemoglobin, performed following standard quality-control procedures.
Change from baseline Glycated Hemoglobin (HbA1c) at 12 months | 12 months
  Venous blood samples will be collected at morning between 7-9 a.m. for the analysis of Glycated Hemoglobin, performed following standard quality-control procedures.

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Zurlo, MD, Principal Investigator — University of Padova

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alawad AO, Merghani TH, Ballal MA. Resting metabolic rate in obese diabetic and obese non-diabetic subjects and its relation to glycaemic control. BMC Res Notes. 2013 Sep 26;6:382. doi: 10.1186/1756-0500-6-382. PMID 24070224
- [Background] Stevenson RW, Parsons JA, Alberti KG. Effect of intraportal and peripheral insulin on glucose turnover and recycling in diabetic dogs. Am J Physiol. 1983 Feb;244(2):E190-5. doi: 10.1152/ajpendo.1983.244.2.E190. PMID 6337503
- [Background] Zawadzki JK, Wolfe RR, Mott DM, Lillioja S, Howard BV, Bogardus C. Increased rate of Cori cycle in obese subjects with NIDDM and effect of weight reduction. Diabetes. 1988 Feb;37(2):154-9. doi: 10.2337/diab.37.2.154. PMID 3391340
- [Background] Piaggi P, Thearle MS, Bogardus C, Krakoff J. Fasting hyperglycemia predicts lower rates of weight gain by increased energy expenditure and fat oxidation rate. J Clin Endocrinol Metab. 2015 Mar;100(3):1078-87. doi: 10.1210/jc.2014-3582. Epub 2015 Jan 5. PMID 25559400
- [Background] Araiza P, Hewes H, Gashetewa C, Vella CA, Burge MR. Efficacy of a pedometer-based physical activity program on parameters of diabetes control in type 2 diabetes mellitus. Metabolism. 2006 Oct;55(10):1382-7. doi: 10.1016/j.metabol.2006.06.009. PMID 16979410
- [Background] Jennings AE, Alberga A, Sigal RJ, Jay O, Boule NG, Kenny GP. The effect of exercise training on resting metabolic rate in type 2 diabetes mellitus. Med Sci Sports Exerc. 2009 Aug;41(8):1558-65. doi: 10.1249/MSS.0b013e31819d6a6f. PMID 19568205
- [Background] Mourier A, Gautier JF, De Kerviler E, Bigard AX, Villette JM, Garnier JP, Duvallet A, Guezennec CY, Cathelineau G. Mobilization of visceral adipose tissue related to the improvement in insulin sensitivity in response to physical training in NIDDM. Effects of branched-chain amino acid supplements. Diabetes Care. 1997 Mar;20(3):385-91. doi: 10.2337/diacare.20.3.385. PMID 9051392
- [Background] Karstoft K, Brinklov CF, Thorsen IK, Nielsen JS, Ried-Larsen M. Resting Metabolic Rate Does Not Change in Response to Different Types of Training in Subjects with Type 2 Diabetes. Front Endocrinol (Lausanne). 2017 Jun 13;8:132. doi: 10.3389/fendo.2017.00132. eCollection 2017. PMID 28659869
- [Derived] Zurlo F, Trevisan C, Vitturi N, Ravussin E, Salvo C, Carraro S, Siffi M, Iob I, Saller A, Previato L, Sergi G, de Kreutzenberg S, Maran A, Avogaro A. One-year caloric restriction and 12-week exercise training intervention in obese adults with type 2 diabetes: emphasis on metabolic control and resting metabolic rate. J Endocrinol Invest. 2019 Dec;42(12):1497-1507. doi: 10.1007/s40618-019-01090-x. Epub 2019 Jul 29. PMID 31359403